CLINICAL TRIAL: NCT03050008
Title: Randomized, Controlled Trial in Patients With Senile Cataract to Evaluate the Efficacy of Ultrasound-free Femtosecond Laser (FLACS) Cataract Surgery (USFREE), Compared to Traditional Phacoemulsification Surgery Using Ultrasound.
Brief Title: Efficacy of FLACS USFREE Compared to Traditional Surgery Using Ultrasound.
Acronym: USFREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alfredo Tranjan Centro Oftalmologico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USFREE
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Senile Cataract; Cataract
Keywords: Cataract Surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FLACS USFREE (Other): Cataract Surgery with Femtosecond Laser Without Ultrasound
  Interventions: Other: FLACS USFREE
- Traditional Surgery (Other): Traditional phacoemulsification cataract surgery using ultrasound
  Interventions: Other: Traditional Surgery

INTERVENTIONS:
Other: FLACS USFREE — Cataract Surgery with Femtosecond Laser Without Ultrasound
  Arms: FLACS USFREE
Other: Traditional Surgery — Traditional phacoemulsification cataract surgery using ultrasound.
  Arms: Traditional Surgery

SUMMARY:
Despite the advantages already demonstrated by FLACS, these surgeries still require ultrasonic devices for fragmentation of the lens. The ultrasonic energy used during phacoemulsification may induce complications such as reduction of endothelial cells and corneal edema. In this sense, it would be beneficial to develop surgical techniques that eliminate the need for ultrasound. The group of surgeons of Alfredo Tranjan Ophthalmic Center, recently developed a surgical technique of cataract that optimizes the use of the laser, eliminating the need for ultrasound during the surgical procedure. Thus, the crystalline fragmentation process does not involve ultrasound being performed by the laser itself. It is expected that this procedure will reduce the complexity of cataract surgery, and be safer in terms of potential corneal lesions. The present study intends to evaluate the benefit and safety of FLACS without use of ultrasound (USFREE), compared to traditional phacoemulsification surgery using ultrasound in patients with senile cataract. In this sense, it is intended to primarily compare the volume of balanced saline solution (BSS) between surgeries.

DETAILED DESCRIPTION:
Study hypothesis:

In cataract surgery, the FLACS USFREE technique is not inferior to the traditional phacoemulsification technique using ultrasound.

Primary Objective:

To compare non-use ultrasound FLACS (USFREE) versus traditional phacoemulsification surgery using ultrasound in eyes undergoing cataract surgery relative to the volume of BSS measured during surgery.

Secondary objective (s):

* To compare cumulative dissipated energy (CDE) used between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound.
* Compare eyes submitted to FLACS USFREE versus traditional phacoemulsification surgery using ultrasound, relative to phacoemulsification time.
* Comparing eyes subjected to FLACS USFREE versus traditional phacoemulsification surgery using ultrasound 1, 7 and 30 days after surgery, for the following parameters:

  * Endothelial cell count.
  * Visual acuity.
  * Corneal topography.
  * The corneal pachymetry.
  * Intraocular pressure.
* Compare the safety profile of FLACS USFREE versus phacoemulsification surgery with ultrasound.

Study design:

Interventional, randomized, open and controlled study.

Study participants will be divided into 2 groups (FLACS without ultrasound and traditional phacoemulsification with ultrasound) and the following visits will be conducted:

* Visit -1 (pre-operative visit - day -30 to day -1 of surgery). Assessment in both eyes. If the two eyes of the research participant are eligible for the study, the eye with the least visual acuity that is designated by O1 will be selected and operated first. The second operated eye will be designated O2.
* Visit 0 (O1 surgery).
* Visit 1 (day 1 [+ 2 days] after O1 surgery).
* Visit 2 (day 7 [± 2 days] after O1 surgery).
* Visit 3 (day 30 [± 2 days] after O1 surgery).

Research participants with the second eligible eye (O2) will further perform the following assessments:

* Visit 4 (O2 surgery, which will occur on the same day of Visit 3 [+ 45 days]).
* Visit 5 (day 1 [± 2 days] after O2 surgery).
* Visit 6 (day 7 [± 2 days] after O2 surgery).
* Visit 7 (day 30 [± 2 days] after O2 surgery). Randomization process The included study participants will be allocated to one of the 2 treatment groups through computer-generated randomization (1: 1 randomization). In research participants with both eyes eligible, the surgical procedure will always be the same for both eyes.

Previously randomized and operated trial participants may not be randomized again in the study.

Concealment process:

This is an open study with no concealment procedures.

Inclusion criteria:

* Male or female gender.
* Age between 40 and 80 years (inclusive).
* Diagnosis of senile type cataract, characterized as grade II nuclear (opacity according to Lens opacities classification system II [LOCS II]), in at least 1 of the eyes.
* Obtaining the informed consent form signed by the research participant and / or legal representative.

Exclusion Criteria:

Research participants or eyes should be excluded in the presence of at least one of the following criteria:

* Cataract of degree other than II (LOCS II).
* Diabetes mellitus.
* History or presence of another ocular pathology.
* History of laser treatment (retinal or iriane).
* History of previous intraocular surgery.
* Endothelial cell count <1500 cells / mm2.
* Corneal thickness> 700 μm.
* Dilated pupil with a diameter <7.0 mm.
* Depth of the anterior chamber <2.5 mm.
* Contraindications for cataract surgery, including:Active proliferative diabetic retinopathy; Rubeosis iridis and / or neovascular glaucoma; Microphthalmia; Buftalmia; The anterior uveitis; The cornea gutatta; Glaucoma; Retinal detachment.
* Other systemic or concomitant diseases that, in the opinion of the investigator, prevent the surgery from being performed or can significantly bias the results.
* Female research participant pregnant or not adhering to appropriate contraceptive measures including abstinence, hormonal contraceptives, diaphragm or condom with spermicide, intrauterine device and surgical sterilization.

Discontinuation criteria (if applicable):

* Withdrawal of consent.
* In case of death.
* Loss of follow-up before the end of the study.
* Greater protocol violation.
* Research participants who do not comply with protocol requirements.
* Any clinical condition or adverse event that, at the discretion of the investigator, impedes the continuation of the research participant in the protocol.

Expected number of eyes: 53 operated eyes per group (106 eyes in total).

Expected number of research centers:

A research center (Alfredo Tranjan Ophthalmological Center).

Selection of research participants:

Research participants followed in the research center (Alfredo Tranjan Ophthalmological Center) and indicated for cataract surgery.

Study Procedures:

Study data will be collected after obtaining the free and informed consent term. Data will be collected for questions to the research participant, consultation of their clinical records and laboratory tests and ocular tests. Surgical data will be obtained during the perioperative period.

Data collection will take place at the research center (Alfredo Tranjan Ophthalmological Center).

Data collected

* Evaluation of the eligibility criteria and signing of the free and informed consent form.
* Socio-demographic data: gender, date of birth.
* Medical history: Identification of the affected eye (s) and Date of diagnosis of cataract in each eye.
* Comorbidities and history of ocular and non-ocular surgeries.
* Non-pharmacological medications and treatments performed at the time of evaluation. Treatments received up to 3 months before the entry of the research participant will be registered.
* Urine test for detection of human chorionic gonadotrophin.
* Retinal mapping in both eyes: observation of the fundus of the eye by a retinal surgeon (the same throughout the study) with Volk 20D magnifying glass to study vessels, optic nerve, macula and retina. Data collected included absence or presence (and specification) of ocular pathology.
* Eye parameters in both eyes

  * Biometrics(Crystalline thickness (mm), Axial length of the eye (mm) and White to white corneal diameter (mm))
  * Endothelial cell count.
  * The corneal pachymetry.
  * Corneal topography.
  * Intraocular pressure.
  * Visual acuity.
* Confirmation of eligibility criteria.
* Randomization of the research participant (USFREE FLACS surgery or standard surgery).
* Volume of saline solution used during surgery.
* Start time and end of surgery.
* Phacoemulsification duration.
* CDE.
* Occurrences during surgery (complications of surgery, adaptations in the procedure).
* Adverse events (other than complications of surgery) since the last evaluation
* Changes in medications and pharmacological treatments concomitant since the last visit.
* Occurrence of adverse events.
* Changes in medications and pharmacological treatments concomitant since the last visit.
* Retinal mapping: absence or presence (and specification) of ocular pathology.

For discontinuing research participants, the primary reason for discontinuation and date of last contact within the study should be collected. Information on adverse events and changes in concomitant treatment that have occurred until discontinuation should also be obtained.

Primary outcome:

- BSS volume difference observed between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery.

Secondary Outcomes:

* Difference in CDE between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery.
* Difference in time (in seconds) of phacoemulsification during surgery, between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery.
* Difference in endothelial cell counts 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound.
* Difference in visual acuity presented 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound.
* Difference in visual acuity with better correction 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery.
* Difference in corneal topography 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound.
* Difference in corneal pachymetry 1, 7 and 30 days after cataract surgery, between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery.
* Difference in intraocular pressure 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery.
* Incidence of adverse events during the study period among study participants submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound.

Statistical methods

Descriptive analyzes:

For the continuous parameters the mean, standard deviation, median, minimum and maximum are given. For the categorical parameters, the cell frequencies and the percentage of research participants in each category will be given.

Primary outcome:

The BSS volume will be summarized using descriptive statistics per surgery group.

The comparison of BSS volume between groups will be determined with a 95% confidence interval, which will be estimated using the analysis of covariance with BSS volume immediately after surgery as the dependent variable, type of surgery as factor and covariables If there are statistical and clinically relevant differences between the two groups regarding their basal characteristics (eg age).

Generalized models will also be used, if applicable.

Other comparative analyzes:

* Time-to-event variables will be compared between groups using the logrank test for comparison of Kaplan-Meier curves.
* Quantitative variables will be compared between groups using the t-test for independent samples, or Mann-Whitney test in case of non-normal distribution.

The level of significance assumed in inferential analyzes will be 0.05. Inferential analysis will be bilaterial.

The data will be analyzed using SAS® Software (version 9.4; SAS Institute Inc, Cary, USA).

Duration of the study:

7 months from the beginning of the recruitment to the completion of the follow-up of the last research participant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of senile cataract, characterized as grade II nuclear (opacity according to Lens opacities classification system II [LOCS II]), in at least 1 of the eyes.
* Obtaining the informed consent form signed by the research participant and / or legal representative.

Exclusion Criteria:

* Cataract of degree other than II (LOCS II).
* Diabetes mellitus.
* History or presence of other ocular pathology.
* History of laser treatment (retinal or iriane).
* History of previous intraocular surgery.
* Endothelial cell count <1500 cells / mm2.
* Corneal thickness> 700 μm.
* Dilated pupil with a diameter of <7.0 mm.
* Depth of the anterior chamber <2.5 mm.
* Contraindications for cataract surgery, including: Active proliferative diabetic retinopathy; Rubeosis iridis and / or neovascular glaucoma; Microphthalmia Buftalmia; The anterior uveitis; The cornea gutatta; Glaucoma; Retinal detachment; Other systemic or concomitant diseases that, in the opinion of the investigator, prevent the surgery from being performed or can significantly bias the results.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Difference in BSS volume observed between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery. | time of surgery
  Difference in BSS (balanced saline solution) volume observed between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery.
  The volume of BSS will be measured during surgery in mL, the sum of the BSS volume observed will be compared between the 2 groups. This volume will be monitored and measured by the Centurion® phacoemulsification device.

SECONDARY OUTCOMES:
Difference in CDE between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery. | time of surgery
  Cumulative dissipated energy is an estimate of the energy used at the incision site during cataract removal and is measured automatically by the Centurion® device in% -seconds. Lower value reflects less energy used, being considered more favorable for the safety of the corneal endothelium.
  For surgeries that occurred according to the first version of this protocol (03-Nov-2015) the CDE data contained in the source documents will be used, , since this is a data already collected during both procedures.
Difference in time (in seconds) of phacoemulsification during surgery, between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery. | time of surgery
  Phacoemulsification time is measured automatically by Centurion®, and expressed in minutes and seconds.
Difference in endothelial cell counts 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound. | Within 30 days after surgery
  The endothelial cell count will be performed in each eye at V1, V1, V2 and V3 (and V5, V6 and V7 for O2) using SP02® specular microscope (CSO, Italy).
Difference in visual acuity presented 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery. | Within 30 days after surgery
  Difference in visual acuity presented 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery.
Difference in visual acuity with best correction 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery. | Within 30 days after surgery
  The visual acuity presented and best corrected will be measured in V-1, V1, V2 and V3 for each eye (and V5, V6 and V7 for O2).
  Assessment of visual acuity in the distance (4 m) will be performed with the standardized and backlit LogMAR table. All exams for this study will be performed with the same equipment and lighting conditions. Research participants will be asked to read the smaller line whose letters are easily distinguishable. Survey participants will continue to read lines with smaller and smaller letters until the survey participant misses all the letters or can not guess any of them. While the survey participant reads the table, the number of letters read incorrectly will be recorded on each line. In this study, the LogMAR of the presented visual acuity and the visual acuity with better correction will be obtained.
Difference in corneal topography 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery. | Within 30 days after surgery
  Simulated keratometry (Yes K) will be measured in each eye at V-1, V1, V2 and V3 (and V5, V6 and V7 for O2) using the Pentacam® system (OCULUS, WA, USA). The Pentacam® system will use a rotating Scheimpflug camera to produce a three-dimensional analysis of the anterior segment of the cornea. A Sim K will be obtained by averaging the power of the anterior surface of the cornea along a 3 mm center ring, measured in diopters (D). In order to minimize bias, measurements will always be made on the same device, with the same operator or their back-up, both with the same training.
Difference in corneal pachymetry 1, 7 and 30 days after cataract surgery, between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery. | Within 30 days after surgery
  In this examination, the pachymeter will be placed in front of the eye to measure the thickness of the cornea, which will be recorded in mm. This analysis will be done in V-1, V1, V2 and V3 (and V5, V6 and V7 for O2). In order to minimize bias, measurements will always be made on the same device, with the same operator or their back-up, both with the same training.
Difference in intraocular pressure 1, 7 and 30 days after cataract surgery between eyes submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound surgery. | Within 30 days after surgery
  Intraocular pressure will be measured in each eye at V-1, V1, V2 and V3 (and V5, V6 and V7 for O2) using the Goldmann aplanation tonometer (Haag-Streit Diagnostics, Switzerland). The intraocular pressure will be measured in mmHg. In order to minimize bias, measurements will always be made on the same device, with the same operator or their back-up, both with the same training.
Incidence of adverse events during the study period among study participants submitted to FLACS USFREE versus traditional phacoemulsification with ultrasound. | Within 30 days after surgery
  Adverse events will be gathered for each eye and each research participant

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Tranjan, MD, Principal Investigator — Alfredo Tranjan Centro Oftalmologico LTDA

IPD SHARING:
Plan to Share IPD: Undecided
Information not yet provided.